CLINICAL TRIAL: NCT02790723
Title: A Phase I Study Evaluating the Safety of Intra-Articular Sc-rAAV2.5IL-1Ra in Subjects With Moderate Osteoarthritis of the Knee
Brief Title: Safety of Intra-Articular Sc-rAAV2.5IL-1Ra in Subjects With Moderate Knee OA
Acronym: AAVIL-1Ra
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher H. Evans, Ph.D., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-007542
Record Dates: First submitted 2016-05-03; First posted 2016-06-06 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose Group (Experimental): Subjects will receive a single intra-articular 2mL injection consisting of 10{11} viral genomes.
  Interventions: Drug: sc-rAAV2.5IL-1Ra
- Medium Dose Group (Experimental): Subjects will receive a single intra-articular 2mL injection consisting of 10{12} viral genomes.
  Interventions: Drug: sc-rAAV2.5IL-1Ra
- High Dose Group (Experimental): Subjects will receive a single intra-articular 2mL injection consisting of 10{13} viral genomes.
  Interventions: Drug: sc-rAAV2.5IL-1Ra

INTERVENTIONS:
Drug: sc-rAAV2.5IL-1Ra — Self-complementing, recombinant AAV carrying IL-1Ra cDNA produced by the Research Institute at Nationwide Children's Hospital.
  Other Names: AAVIL-1Ra; IL-1Ra

SUMMARY:
This study seeks to determine the safety of three different doses of sc-rAAV2.5IL-1Ra delivered by intra-articular injection into one knee joint of patients with moderate OA of the knee.

ELIGIBILITY:
Inclusion Criteria

* Age 18-80 years
* Gender: both males and females
* Target disease: Moderate OA of the knee
* Persistent symptoms, despite standard NSAID
* Absence of clinically significant abnormal values for the following:
* Complete blood count
* Prothrombin Time, Activated partial thromboplastin time
* Blood chemistry (Glucose, Na, K, Cl, CO2, BUN, creatinine, Ca, PO4, magnesium, uric acid)
* Liver function tests (amylase, total bilirubin, alkaline phosphate, GGT, AST, ALT, total protein, albumin)
* Able and willing to return to the Mayo Clinic for follow-up visits, as required by this study
* Able undergo MRI of the knee
* Subjects should be able to give appropriate consent.
* Potential subjects should have failed a three-month trial of a minimum of two conservative therapies before being considered for this trial. These conservative therapies include: activity modification, weight loss, physical therapy, and anti-inflammatory or injection therapy.

Exclusion Criteria

* Pregnant, or currently breast-feeding
* Ongoing infectious disease including HIV, HTLV, hepatitis, syphilis or tuberculosis positive
* Individuals who have OA as part of another syndrome (e.g. Ehler's Danlos, Stickler syndrome, etc.)
* Systemic, rheumatic or inflammatory disease of the knee or chondrocalcinosis, hemochromatosis, inflammatory arthritis, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's knee joint, villonodular synovitis, and synovial chondromatosis.
* Clinically significant cardiovascular, renal, hepatic, endocrine disease, diabetes, cancer, autoimmune diseases; a serious infection or major operation within 30 days of enrollment; a history of untreated psychiatric disease or recent history of alcoholism or drug addiction.
* Currently taking immunosuppressant medications
* Anticipated major surgery during the study period.
* Individuals involved in another interventional protocol, or have been treated under one within the last 3 months.
* Intra-articular therapy in the index knee within the previous 3 months.
* Surgery to the target knee within 6 months prior to screening.
* Surgery to other weight bearing joints if it will interfere with knee assessments
* Prior articular transplant procedures
* Orthopedic hardware or implantable devices in the index knee
* Prior reconstruction surgery to the target knee within 12 months
* X-ray findings of acute fractures
* Known severe loss of bone density, and/or severe bone or joint deformity in the target knee.
* Significant target knee infection or overlying skin disorder/infection within the previous 6 months prior to study enrollment
* Require cane or other assistive device for walking
* Symptomatic OA of the hips, spine or ankle if it would interfere with the evaluation of the target knee,
* History of documented nerve damage in the affected limb, or vascular insufficiency,
* Condition requiring use of systemic steroids,
* Coagulation disorder.
* Patients with unstable knees
* Temperature above 99.5o F.
* Identification as a member of a vulnerable population.
* BMI greater than 40.
* History of allergy to local anesthetics
* Currently taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within the 3 months prior to entry in the study.
* Any illness or condition which, in the investigators' judgement will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing severe adverse events. | 53 weeks
  Assess the local and systemic safety of three different doses of sc-rAAV2.5IL-1Ra delivered by intra-articular injection into one knee joint of patients with moderate OA of the knee.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H. Evans, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans CH, Ghivizzani SC, Robbins PD. Osteoarthritis Gene Therapy: A 30-Year Journey From Concept to Clinical Trials. J Orthop Res. 2026 Feb;44(2). doi: 10.1002/jor.70141. PMID 41607103
- [Derived] Evans CH, Ghivizzani SC, Robbins PD. The 2024 OREF Clinical Research Award: Progress Toward a Gene Therapy for Arthritis. J Am Acad Orthop Surg. 2024 Dec 1;32(23):1052-1060. doi: 10.5435/JAAOS-D-24-00831. Epub 2024 Oct 17. PMID 39284030
- [Derived] 2022 AMSSM Rising With Research Presentations. Clin J Sport Med. 2022 Mar 1;32(2):168-176. doi: 10.1097/JSM.0000000000001014. No abstract available. PMID 35234744
- [Derived] 2021 AMSSM Oral Research Poster Presentations. Clin J Sport Med. 2021 Mar 1;31(2):185-221. doi: 10.1097/JSM.0000000000000914. No abstract available. PMID 33647918
- [Derived] Mehta S, He T, Bajpayee AG. Recent advances in targeted drug delivery for treatment of osteoarthritis. Curr Opin Rheumatol. 2021 Jan;33(1):94-109. doi: 10.1097/BOR.0000000000000761. PMID 33229973
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials